CLINICAL TRIAL: NCT00144261
Title: An Open-label, Non-randomized, Single-arm Study, to Investigate the Mechanism(s) by Which Nevirapine Increases Plasma High Density Lipoproteins Concentration in HIV+ Subjects Treated With VIRAMUNE® Tablets
Brief Title: An Open-label, Non-randomized, Single-arm Study to Investigate the Mechanism(s) by Which Nevirapine Increases Plasma HDL in HIV+ Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: 1100.1426
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections; Metabolism, Lipids
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

INTERVENTIONS:
Drug: nevirapine

SUMMARY:
1. In order to obtain further insight as to how NVP affects HDL metabolism, the in vivo kinetics of the HDL apolipoprotein, Apo A-1, before and 6 weeks after initiation of NVP containing treatment were evaluated. In addition, the activity of the key enzymes related to HDL metabolism were assessed.

   [ Designated as safety issue: No ]
2. In order to determine the relevance of the HDL increase in decreasing cardiovascular risk in HIV-positive subjects we evaluated endothelial function (FMD) as a surrogate marker for cardiovascular disease in patients.

[ Designated as safety issue: No ]

ELIGIBILITY:
Inclusion Criteria:

Patients will be included when they meet the following criteria:

1. 18 years of age or older.
2. Ability and willingness to provide signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.
3. Patients on stable therapy with Trizivir only (or its equivalent component drugs), for at least 6 months prior to screening.
4. Patients with plasma HIV-1-RNA <=50 copies/mL documented on at least two occasions within 6 months prior to enrollment.
5. Documentation of plasma HIV-1 RNA of <=50 copies/mL for >=6 months while on Trizivir without other antiretroviral agent. Documentation will include dates and results of all viral load testing from the previous six months.
6. Ability and willingness to complete the study.

Exclusion Criteria:

Patients will not be included when they meet one or more of the following criteria:

1. Previous exposure to NNRTI drugs.
2. Documented diabetes mellitus.
3. Documented hypertension (systolic >155 mmHg and/or diastolic >95 mmHg).
4. Fasting hypertriglyceridemia (>5.6 mmol/L or 500 mg/dl).
5. Use of lipid-lowering medication during the 90 days prior to study enrollment.
6. Chronic active hepatitis B and/or C infection by history.
7. Anemia (Hb <7.0 mmol/l or 11 g/dl hematocrit <32%).
8. Active opportunistic infection or neoplasm within 3 months prior to screening visit with the exception of cutaneous Kaposi's sarcoma without evidence of progressive disease.
9. Any history of cardiovascular disease (infarction, heart failure, peripheral vascular disease, cerebrovascular disease).
10. Hepatic, renal or thyroid abnormalities, as determined significant by the Principal Investigator.
11. Pregnancy or lactation.
12. Active anticoagulation therapy (coumarin derivates, heparin).
13. History of HIV-2 infection.
14. Female patients with CD4 counts >250 cells/mm3.
15. Male patients with CD4 counts >400 cells/mm3. Others which can not be listed here.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11-01 (Actual); Primary Completion 2006-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage change of fractional synthetic rate (FSR) of Apo A-1 | after 6 weeks of treatment
Percentage change of flow mediated dilatation (FMD) | after 6 and 24 weeks of treatment

SECONDARY OUTCOMES:
Percentage change in the proteins involved in HDL metabolism | after 6 and 24 weeks of treatment
The percentage change in plasma levels of lipoproteins in the fasting lipid panel (TC, LDL, HDL, TG) from Week 0 (baseline) to 6 and 24 weeks of treatment with NVP-based antiretroviral therapy | from week 0 to 6, and 24 weeks of treatment
The percentage change in activity (and/or mass) of the constituents of the lipid enzymes panel from Week 0 to 24 weeks of NVP-based antiretroviral therapy | from week 0 to 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Netherlands (2):
  - 1100.1426.01 Academic Medical Centre, Amsterdam
  - 1100.1426.02 Onze Lieve Vrouwe Gasthuis, Amsterdam
- 1100.1426.44001 Boehringer Ingelheim Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/19667106